CLINICAL TRIAL: NCT00856700
Title: Effect of GLP-1 on Endothelial Function and Glucose Uptake in Patients With Metabolic Syndrome
Brief Title: Glucagon-like Peptide 1 (GLP-1) and Endothelial Dysfunction in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Manfredi Tesauro, Associate Professor of Internal Medicine, University of Rome Tor Vergata
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 144/08
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome
Keywords: GLP-1; Endothelial Function; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Incretins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GLP-1 infusion (Experimental): Patients with metabolic syndrome
  Interventions: Drug: GLP-1 infusion

INTERVENTIONS:
Drug: GLP-1 infusion — Participants will receive intraarterial infusion of GLP-1 (20 pmol/ml solution) for 100 min.
  Other Names: Incretins

SUMMARY:
Glucagon-like peptide 1 (GLP-1) is an intestinal peptide hormone secreted in a nutrient-dependent manner that stimulates the pancreatic beta cells to secrete more insulin in response to the same amount of blood glucose. In patients with Type 2 diabetes, GLP-1 secretion is lower than normal, thus suggesting that the hormone may contribute to the pathogenesis of the disease. Whether infusion of GLP-1 affects endothelial function and glucose uptake in humans has never been investigated. In the current proposal, the investigators hypothesize that GLP-1 administration might ameliorate endothelial dysfunction in patients with metabolic syndrome. To test this hypothesis, the investigators will evaluate the acute effects of GLP-1 in the forearm circulation of patients with metabolic syndrome during local hyperinsulinemia by use of the forearm perfusion technique.

DETAILED DESCRIPTION:
Subjects meeting the entrance criteria will be studied in a quiet room with a temperature of approximately 22°C. While the participants are supine, a 20-gauge Teflon catheter will be inserted into the brachial artery of the nondominant arm under local anesthesia. This arm will be slightly elevated above the level of the heart, and a mercury-filled Silastic strain gauge will be placed on the widest part of the forearm. The strain gauge will be connected to a plethysmography calibrated to measure the percent change in volume; the plethysmograph in turn will be connected to a chart recorder to record the forearm flow measurements. For each measurement, a cuff placed on the upper arm will be inflated to 40 mmHg with a rapid cuff inflator to occlude venous outflow from the extremity. A wrist cuff will be inflated to suprasystolic pressures l min before each measurement to exclude the hand circulation. Flow measurements will be recorded for approximately 7 seconds every 15 seconds; 7 readings will be obtained for each value.

The intraarterial catheter will be connected by a 3-way stopcock to both a pressure transducer (to measure intraarterial blood pressure) and an infusion pump. Saline or drugs then will be infused at the rate of 0.5-1ml per minute. Another 20-gauge Teflon catheter will be inserted in a homolateral antecubital vein for blood sampling.

To assess the effects of GLP-1 on insulin stimulated vasodilation, after the forearm will be instrumented, patients with metabolic syndrome will receive intraarterial infusion of saline for 15 minutes; blood samples will be collected and baseline flow will be measured. Then infusion of regular insulin (Humulin, Eli Lilly, Indianapolis, IN; 0.1 mU per kg of body weight per minute) will be started. Next, forearm blood flow will be measured after infusion of Ach, a vasodilator whose effect is predominantly related to nitric oxide (NO), and sodium nitroprusside (SNP), an exogenous NO donor.

After 20 min of insulin infusion, another baseline measurement will be obtained and continuous intraarterial infusion of GLP-1 will be started at 20 pmol/min infusion rate. This dose has been chosen in order to achieve intravascular GLP-1 concentrations within the infused forearm in a range (approximately 0.50 pmol/mL) previously shown effective to improve insulin sensitivity. GLP-1 infusion will be continued for 60 minutes, and forearm blood flow will be measured every 30 minutes; venous blood samples will be obtained at the end of this infusion period. Then, while maintaining GLP-1 infusion unchanged, dose-response curves to ACh and SNP will be repeated, at the same doses and following the same protocol as before.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy individuals aged between 20 and 60 years
* Must satisfy 3 out of the 5 listed criteria for the diagnosis of the metabolic syndrome (ATP III) will be included

Exclusion Criteria:

* Pregnancy
* Liver disease
* Pulmonary disease
* Renal insufficiency
* Coronary heart disease
* Heart failure
* Peripheral vascular disease
* Coagulopathy
* Any disease predisposing to vasculitis or Raynaud's phenomenon
* Bleeding disorders
* Kidney stones
* Platelet count < 150,000/ml blood
* Prothrombin time/partial thromboplastin time (PT/PTT) > 1 second above the normal range, and positive tests for HIV, or hepatitis B or C
* Subjects who are taking any kind of medication will not be included in this study; therefore, antihypertensive and/or lipid-lowering drugs will be discontinued at least 2 weeks before enrollment into this study
* All subjects will be told to refrain from alcohol, beverages containing caffeine, or smoking for at least 24 hours before the study is performed

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent vasodilation capacity | 60 minutes

SECONDARY OUTCOMES:
Insulin-mediated glucose uptake | 100 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Manfredi Tesauro, MD, Principal Investigator — Internal Medicine Department, Tor Vergata University, Rome
Locations (1):
- Tor Vergata University, Rome, Italy

REFERENCES:
- [Background] Tesauro M, Schinzari F, Rovella V, Melina D, Mores N, Barini A, Mettimano M, Lauro D, Iantorno M, Quon MJ, Cardillo C. Tumor necrosis factor-alpha antagonism improves vasodilation during hyperinsulinemia in metabolic syndrome. Diabetes Care. 2008 Jul;31(7):1439-41. doi: 10.2337/dc08-0219. Epub 2008 Apr 4. PMID 18390795
- [Background] Tesauro M, Schinzari F, Iantorno M, Rizza S, Melina D, Lauro D, Cardillo C. Ghrelin improves endothelial function in patients with metabolic syndrome. Circulation. 2005 Nov 8;112(19):2986-92. doi: 10.1161/CIRCULATIONAHA.105.553883. Epub 2005 Oct 31. PMID 16260640
- [Background] Zander M, Madsbad S, Madsen JL, Holst JJ. Effect of 6-week course of glucagon-like peptide 1 on glycaemic control, insulin sensitivity, and beta-cell function in type 2 diabetes: a parallel-group study. Lancet. 2002 Mar 9;359(9309):824-30. doi: 10.1016/S0140-6736(02)07952-7. PMID 11897280
- [Background] Toft-Nielsen MB, Madsbad S, Holst JJ. Continuous subcutaneous infusion of glucagon-like peptide 1 lowers plasma glucose and reduces appetite in type 2 diabetic patients. Diabetes Care. 1999 Jul;22(7):1137-43. doi: 10.2337/diacare.22.7.1137. PMID 10388979
- [Derived] Tesauro M, Schinzari F, Adamo A, Rovella V, Martini F, Mores N, Barini A, Pitocco D, Ghirlanda G, Lauro D, Campia U, Cardillo C. Effects of GLP-1 on forearm vasodilator function and glucose disposal during hyperinsulinemia in the metabolic syndrome. Diabetes Care. 2013 Mar;36(3):683-9. doi: 10.2337/dc12-0763. Epub 2012 Oct 15. PMID 23069838